CLINICAL TRIAL: NCT04071639
Title: Non-randomized Control Clinical Trial to Evaluate the Efficacy and Safety of Symptomatic Drug Therapy for Mild to Moderate Huntington's Disease Patients
Brief Title: Symptomatic Therapy for Patients With Huntington's Disease
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019238
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2021-04-02 (Actual); Status verified 2021-03

CONDITIONS: Huntington Disease
MeSH Terms: conditions — Huntington Disease | interventions — Haloperidol; Risperidone; Sertraline; Tablets; idebenone; deutetrabenazine

STUDY DESIGN:
Intervention Model Description: Case group use Deutetrabenazine，Risperidone，Zoloft and Idebenone(depending on demand and symptom).
  Control group use Haloperidol，Risperidone，Zoloft and Idebenone(depending on demand and symptom).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Mild to moderate HD patients receive medicine treatment with different doses of Deutetrabenazine(Austedo), Risperidone, Zoloft+Idebenone, according to their symptoms. The mode of administration is oral. Capsules will be swallowed whole with water. Zoloft should be taken 50mg once in the morning and Risperidone 1mg once at night. Deutetrabenazine(Austedo) should be taken 6mg once a day, or increase dose according to AUSTEDO® tablets Prescribing Information. Idebenone should be taken 30mg three times a day. Study drug can be taken irrespective of meals. Duration:5 years.
  Interventions: Drug: Risperidone 1Mg Tab; Drug: Zoloft 50Mg Tablet; Drug: Idebenone; Drug: Deutetrabenazine Oral Tablet [Austedo]
- Group 2 (Experimental): Mild to moderate HD patients receive medicine treatment with different doses of Haloperidol, Risperidone, Zoloft+Idebenone, according to their symptoms. The mode of administration is oral. Capsules will be swallowed whole with water. Haloperidol should be taken 0.5mg~1mg three times a day. The administration of Zoloft, Risperidone and Idebenone are same as group 1. Study drug can be taken irrespective of meals. Duration:5 years.
  Interventions: Drug: Haloperidol 2Mg Tab; Drug: Risperidone 1Mg Tab; Drug: Zoloft 50Mg Tablet; Drug: Idebenone

INTERVENTIONS:
Drug: Haloperidol 2Mg Tab — Haloperidol take 0.5mg~2mg three time a day.
  Other Names: Haloperidol Tables, H31021234
  Arms: Group 2
Drug: Risperidone 1Mg Tab — Risperidone take 1mg once at night.
  Other Names: Risperidone, H20010309
Drug: Zoloft 50Mg Tablet — Zoloft take 50mg once in the morning.
  Other Names: Sertraline Hydrochloride Tablets, H10980141
Drug: Idebenone — Idebebone take 30mg three times a day.
  Other Names: Idebenone,H10970363
Drug: Deutetrabenazine Oral Tablet [Austedo] — The recommended starting dose of Austedo is 6 mg administered orally once daily, and dose may be increased at weekly intervals in increments of 6 mg per day to a maximum recommended daily dosage of 48 mg.
  Other Names: Deutetrabenazine
  Arms: Group 1

SUMMARY:
Based on the previous symptomatic treatment of Chinese HD patients, this study intends to further optimize the treatment regimen of Chinese HD patients so as to further improve the prognosis of patients.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate symptomatic treatment regimen efficacy based on different disease stages. We previously used symptomatic treatment on Chinese HD patients and most of them got improved both in the motor symptoms and life quality. So this study intends to further optimize the treatment regimen, and set a control group to further evaluate the treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Genetic diagnosis of Huntington's disease
2. Symptomatic patients with Huntington's disease
3. Disease duration less than 5 years -

Exclusion Criteria:

(1) Movement disorder due to other definite causes instead of Huntington's disease (2) Severe Lung, kidney or liver disease (3) Neoplastic Disease

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-03-12 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
The Unified Huntington's Disease Rating Scale | Five years
  The Unified Huntington's Disease Rating Scale consist of four subscales, including motor(0-124), MMSE (0-30), psychiatric (0-176), and functional domains(1-13). Four subscale scores are summed to compute a total score. Higher motor and psychiatric scores represent worse outcomes but higher MMSE score and functional scores indicate good outcome.

SECONDARY OUTCOMES:
Brain MRI | Five years
  Brain MRI is used to assess the atrophy of caudate nucleus and cortex in HD patients

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Ying Wu, Study Chair — Second affiliated Hospital, Zhejiang University School of Medicine
Locations (1):
- Second Affiliated Hospital,Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No